CLINICAL TRIAL: NCT05097508
Title: Effect of Atracurium and Rocuronium on the State and Response Entropy During Isoflurane Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noran Essam Mohamed Hassanien, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Noran Hassanien
Record Dates: First submitted 2021-10-05; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Entropy Device and How Will Muscle Relaxants Affect it
Keywords: entropy, atracurium, rocuronium
MeSH Terms: interventions — Atracurium; Rocuronium; Neuromuscular Monitoring

STUDY DESIGN:
Intervention Model Description: * Group A: Patients will receive Atracurium.
  * Group R: Patients will receive rocuronium.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Patients will receive Atracurium. (Experimental): Baseline RE and SE will be recorded. Anesthesia will be induced by propofol (dose 2-3 mg/kg) and fentanyl as analgesia (dose 1-2 mg/kg). Tracheal intubation will be facilitated with atracurium (dose 0.5 mg/kg) after an acceleromyography count of 0. Anesthesia will be maintained with isoflurane in an air-O2 mixture (FiO2 0.6, 2 L/min). Mechanical ventilation will be maintained at a tidal volume of 5-7 ml/kg. Ventilator frequency will be adjusted for maintenance of an ETCO2 of 35-40 mmHg. After equilibrium for 30 minutes SE, RE and the difference between them will be recorded at MAC 0.8 and MAC 1 at two levels of muscle relaxation assessed by TOF value of 50% and 100%. Atracurium (dose 0.005-0.01 mg/kg/min) will be administered as a continuous IV infusion adjusted until 50% and 100% depression of T1 ( first twitch by acceleromyography) will be observed. The entire experiment ended before the start of surgery.
  Interventions: Drug: Atracurium Besylate; Device: Entropy; Device: train of four
- Group R: Patients will receive rocuronium. (Experimental): Baseline RE and SE will be recorded. Anesthesia will be induced by propofol (dose 2-3 mg/kg) and fentanyl as analgesia (dose 1-2 mg/kg). Tracheal intubation will be facilitated with rocuronium (dose 0.6 mg/kg) after an acceleromyography count of 0. Anesthesia will be maintained with isoflurane in an air-O2 mixture (FiO2 0.6, 2 L/min). Mechanical ventilation will be maintained at a tidal volume of 5-7 ml/kg. Ventilator frequency will be adjusted for maintenance of an ETCO2 of 35-40 mmHg. After equilibrium for 30 minutes SE, RE and the difference between them will be recorded at MAC 0.8 and MAC 1 at two levels of muscle relaxation assessed by TOF value of 50% and 100%. Rocuronium (dose 0.01-0.012 mg/kg/min ) will be administered as a continuous IV infusion adjusted until 50% and 100% depression of T1 ( first twitch by acceleromyography) will be observed. The entire experiment ended before the start of surgery.
  Interventions: Drug: Rocuronium Bromide; Device: Entropy; Device: train of four

INTERVENTIONS:
Drug: Atracurium Besylate — Anesthesia will be induced by atracurium (dose 0.5 mg/kg).After equilibrium for 30 minutes SE, RE and the difference between them will be recorded at MAC 0.8 and MAC 1 at two levels of muscle relaxation assessed by TOF value of 50% and 100%. Atracurium (dose 0.005-0.01 mg/kg/min) will be administered as a continuous IV infusion adjusted until 50% and 100% depression of T1 ( first twitch by acceleromyography) will be observed. The entire experiment ended before the start of surgery. In case of hypotension (drop of blood pressure ˃20% of baseline reading), 10-30 mg of ephedrine diluted over 10 ml normal saline 0.9% will be given intravenously by titration according to the blood pressure. In case of bradycardia (heart rate less than 60 beat per minute), when it is associated with hypotension or any signs of impaired perfusion, 0.01 - 0.02 mg/kg of atropine will be given
  Other Names: Tracium
  Arms: Group A: Patients will receive Atracurium.
Drug: Rocuronium Bromide — Anesthesia will be induced by rocuronium (dose 0.6 mg/kg).After equilibrium for 30 minutes SE, RE and the difference between them will be recorded at MAC 0.8 and MAC 1 at two levels of muscle relaxation assessed by TOF value of 50% and 100%. Rocuronium (dose 0.01-0.012 mg/kg/min ) will be administered as a continuous IV infusion adjusted until 50% and 100% depression of T1 ( first twitch by acceleromyography) will be observed. The entire experiment ended before the start of surgery. In case of hypotension (drop of blood pressure ˃20% of baseline reading), 10-30 mg of ephedrine diluted over 10 ml normal saline 0.9% will be given intravenously by titration according to the blood pressure. In case of bradycardia (heart rate less than 60 beat per minute), when it is associated with hypotension or any signs of impaired perfusion, 0.01 - 0.02 mg/kg of atropine will be given.
  Other Names: Esmeron
  Arms: Group R: Patients will receive rocuronium.
Device: Entropy — No premedication will be given. After the patients enter the operating room, a venous cannula will be inserted into a large peripheral vein. Data from routine monitoring, including non-invasive arterial blood pressure, oxygen saturation, and end-tidal oxygen concentration (ETO2) and end-tidal carbon dioxide concentration (ETCO2) will be collected. Neuromuscular blockade will be continuously assessed by acceleromyography using the Train-of-Four-watch SX system , starting when the patients will be unconscious. RE and SE will be monitored using a Datex Ohmeda Entropy Module (M-Entropy) and the Entropy Sensor system.
Device: train of four — After the patients enter the operating room, a venous cannula will be inserted into a large peripheral vein. Data from routine monitoring, including non-invasive arterial blood pressure, oxygen saturation, and end-tidal oxygen concentration (ETO2) and end-tidal carbon dioxide concentration (ETCO2) will be collected. Neuromuscular blockade will be continuously assessed by acceleromyography using the Train-of-Four-watch SX system, starting when the patients will be unconscious. RE and SE will be monitored using a Datex Ohmeda Entropy Module (M-Entropy) and the Entropy Sensor system.

SUMMARY:
Many studies have explored the effects of inhalation anesthetics, intravenous anesthetics, and muscle relaxants on spectral entropy, but most did not monitor the degree of neuromuscular block. In addition, they do not explore the effects of different degrees of neuromuscular blockade on spectral entropy under different concentrations of isoflurane inhalation. Therefore, the present study will evaluate different levels of MAC to quantify the isoflurane concentration, as well as different degrees of neuromuscular blockade

DETAILED DESCRIPTION:
The study will include 40 patients fulfilling the inclusion criteria. They will be randomized into 2 equal groups by a computer generated random numbers table, each consisting of 20 patients, namely group A and group R.

* Group A: Patients will receive Atracurium.
* Group R: Patients will receive rocuronium. No premedication will be given. After the patients enter the operating room, a venous cannula will be inserted into a large peripheral vein. Data from routine monitoring, including non-invasive arterial blood pressure, oxygen saturation, and end-tidal oxygen concentration (ETO2) and end-tidal carbon dioxide concentration (ETCO2) will be collected. Neuromuscular blockade will be continuously assessed by acceleromyography using the Train-of-Four-watch SX system (made in Ireland), starting when the patients will be unconscious. RE and SE will be monitored using a Datex Ohmeda Entropy Module (M-Entropy) and the Entropy Sensor system (made in finland).

Baseline RE and SE will be recorded. Anesthesia will be induced by propofol (dose 2-3 mg/kg) and fentanyl as analgesia (dose 1-2 mg/kg). Tracheal intubation will be facilitated with rocuronium (dose 0.6 mg/kg) /atracurium (dose 0.5 mg/kg) after an acceleromyography count of 0. Anesthesia will be maintained with isoflurane in an air-O2 mixture (FiO2 0.6, 2 L/min). Mechanical ventilation will be maintained at a tidal volume of 5-7 ml/kg. Ventilator frequency will be adjusted for maintenance of an ETCO2 of 35-40 mmHg. After equilibrium for 30 minutes SE, RE and the difference between them will be recorded at MAC 0.8 and MAC 1 at two levels of muscle relaxation assessed by TOF value of 50% and 100%. Rocuronium (dose 0.01-0.012 mg/kg/min ) /atracurium (dose 0.005-0.01 mg/kg/min) will be administered as a continuous IV infusion adjusted until 50% and 100% depression of T1 ( first twitch by acceleromyography) will be observed. The entire experiment ended before the start of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of Anesthesiologists physical status (ASA) I to II.
2. Male patients (to avoid bias between gender).
3. Age between 20-50 years

Exclusion Criteria:

* a. Patients receiving any neuropsychiatric medications. b. Patients undergoing neurosurgical operation. c. Drug addiction. d. Body mass index (BMI) more than or equal to 40.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the impact of different degrees of neuromuscular blockade on SE, RE, and RE-SE difference during isoflurane anesthesia. | 1 year
  to measure effect of atracurium and rocuronium on entropy readings(state,respose and difference between them) during isoflurane anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Noran Hassanien, Principal Investigator — AinShams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collecting IPD will be shared
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year
Access Criteria: anesthesiologist

REFERENCES:
- [Result] Xing Y, Xu D, Xu Y, Chen L, Wang H, Li S. Effects of Neuromuscular Blockages on Entropy Monitoring During Sevoflurane Anesthesia. Med Sci Monit. 2019 Nov 15;25:8610-8617. doi: 10.12659/MSM.917879. PMID 31729355